CLINICAL TRIAL: NCT04261582
Title: Genetics and Genomics of Aspirin Exacerbated Respiratory Disease (AERD)
Acronym: AERD
Status: Suspended | Type: Observational
Why Stopped: On hold due to COVID-19 outbreak
Sponsor: National Jewish Health (Other)
Collaborators: The Scripps Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HS-3200sIRB
Record Dates: First submitted 2019-12-05; First posted 2020-02-10 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Aspirin Exacerbated Respiratory Disease; Aspirin-Sensitive Asthma; Nasal Polyps
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AERD participants: Participants with aspirin exacerbated respiratory disease. Adults with aspirin allergy, nasal polyps and adult-onset severe asthma.
- Healthy controls: Healthy participants that do not have asthma.
- Non-aspirin sensitive asthma participants: Participants with asthma, but that do not have a sensitivity to aspirin.

SUMMARY:
Aspirin Exacerbated Respiratory Disease (AERD) is a relatively homogeneous disease characterized by adult-onset severe asthma, development of non-cancerous growths in the nasal canal (i.e. nasal polyps) and aspirin allergy. The cause of AERD is unknown, although likely results from environmental insults in combination with genetic susceptibility. AERD disease homogeneity increases the possibility of discovering narrowly-defined genetic contributors, and makes it an ideal population to study the genetic and epigenetic changes that cause asthma. Researchers recently discovered that gene expression of epithelial growth and repair (EGR) genes are substantially decreased in bronchial airway epithelial cells of severe asthmatics compared to less severe asthmatics and healthy controls. This new finding indicates that epithelial integrity and related processes may be of primary importance to the development of severe asthma, and potentially the severe asthma subtype, AERD. This finding was later supported in a subsequent lab model, which showed that blocking a central epithelial repair and differentiation gene, human epidermal growth factor receptor 2 (ERBB2), decreased healing time of bronchial epithelial cells after injury. Thus, the objective of the proposed study is to determine whether EGR gene are also down-regulated in AERD, a homogeneous severe asthma subtype. As an extension, the researchers will also determine whether genetic mutations and/or epigenetic changes relate to and potentially explain this down-regulation of EGR genes. Specifically, the researchers plan to obtain gene expression of freshly brushed nasal airway epithelial cells of 140 AERD patients, 70 non-aspirin sensitive asthma patients, and 35 healthy controls, noting that nasal epithelial gene expression has recently been shown to mirror lung epithelial changes in asthmatic airways. Swabbing the nasal canal for epithelial cells allows to evaluate airway epithelial cell gene expression non-invasively. Our experimental design contrasts AERD gene expression profiles against healthy controls, and determines whether EGR genes are depressed in AERD relative to health controls. As a corollary, the researchers look to discover an AERD-specific gene expression profile which may one-day aid in diagnosis and expand current knowledge of disease mechanisms. As an extension, the researchers will correlate gene expression changes, specifically any finding of down-regulated EGR genes, with methylation changes (i.e. epigenetic changes) and genetic mutations.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma
* Physician diagnosis of chronic nasal disease featuring nasal polyps
* Sensitivity to aspirin verified by an aspirin provocative challenge in clinic
* Healthy control participant

Exclusion Criteria:

* Active smoking
* Pregnancy
* History of greater than or equal to 10 pack-years of smoking
* Any significant comorbid conditions that could inadvertently interfere with study results
* Conditions that require bursts of oral corticosteroids
* Other significant lung diseases
* Other disease in the view of the investigator prohibits participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AERD participants, a subtype of severe asthma characterized by inflammation of the nasal cavity, development of non-cancerous growths, and an allergy to aspirin; 35 healthy control participants. Populations will be recruited from clinic visits or clinical research inquiries, all volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of EGR related gene expression in AERD | Through study completion, 3 years
  Researchers will obtain global gene expression of freshly brushed nasal airway epithelial cells of AERD patients, non-aspirin sensitive asthma patients, and healthy patients using nasal swab samples and running RNAseq on the collected cells. Researchers will contrast AERD gene profiles against non-aspirin sensitive asthma patients and healthy patients and determine whether down-regulation of EGR genes is found in AERD.

SECONDARY OUTCOMES:
Relation of EGR gene expression to epigenetic gene methylation | Through study completion, 3 years
  To determine whether whole genome methylation profiling is altered in association with down-regulated EGR genes. Researchers will obtain complementary whole-genome methylation profiles of the study participants and will evaluate whether down-regulated EGR genes in AERD patients are associated with methylation differences by a composite analysis integrating expression and epigenetic data. MethylMix R software program will be used to identify methylation changes associated with gene expression changes. MethylMix integrates DNA methylation from normal and disease samples with matched gene expression. In summary, MethylMix defines hyper and hypomethylated genes by comparing methylation values of disease tissue vs. normal.
Influence of Genetic variation on EGR related gene expression | Through study completion, 3 years
  To determine whether genetic mutations associate with down-regulated EGR gene expression in AERD patients. We will obtain genotypes on these same study participants and evaluate whether down-regulated EGR genes are associated with mutations by a composite analysis integrating expression and genotypes. The Affymetrix genotyping workflow consists of 4 steps; first 3 steps use a set of stand-alone software packages, and the 4th step using R package SNPolisher. Sample QC will be evaluated by Dish-QC statistic, retaining samples with default Dish-QC > 82%. Genotyped samples with a call rate lower than default value of 97% will be excluded. Platewise QC will be evaluated by manually calculating 'Plate Pass Rate' and 'Average Plate Call Rate' statistics, with default cutoff values of 95 and 99%. Genotyping step will be rerun for samples passing quality criteria. SNPolisher will evaluate quality of the signal and classify each SNP probe.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States